CLINICAL TRIAL: NCT04971369
Title: Safety Study of 89Zr-NY001 PET Imaging in Patients With Fibronectin ED-B Positive Solid Tumors
Brief Title: Safety Study of 89Zr-NY001 PET Imaging in Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuxi No. 4 People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Wuxi-4 PH NY001
Record Dates: First submitted 2021-07-20; First posted 2021-07-21 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-NY001 injection (Experimental): Patients will receive a tracer (5 mg, IV) dose of Zr-89 (1.5-2 mCi) labeled NY001 (89Zr-NY001)
  Interventions: Diagnostic Test: 89Zr-NY001

INTERVENTIONS:
Diagnostic Test: 89Zr-NY001 — 89Zr-NY001 injection followed by 89Zr-NY001 PET scan

SUMMARY:
This is a single arm study to evaluate the safety and biodistribution of 89Zr-labeled NY001 (89Zr-NY001) PET imaging in patients with fibronectin ED-B domain positive solid tumors.

DETAILED DESCRIPTION:
After being fully informed about the study and potential risks, all patients giving written informed consent will be evaluated to determine eligibility for study entry. Patients will receive an injection of 89Zr-NY001 and will undergo PET/CT scanning to determine uptake of 89Zr-NY001 in tumor lesions and the whole body.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily signed informed consent;
2. Aged >18, male or female;
3. Patients diagnosed with solid tumors confirmed by histopathology or cytology test;
4. At least two measurable solid lesions has been examined by 18F-FDG PET/CT (RECIST1.1 standard);
5. Patients with biopsy-proven fibronectin ED-B positive;
6. ECOG score ≤ 0~3; Life expectancy of at least 3 months;
7. Women of childbearing age are required to receive serum pregnancy tests, and only those who have a negative pregnancy test for eligible subjects;
8. ALT, AST shall not exceed 3 times of the normal upper limit; Bun, Cr not exceed 1.5 times of the normal upper limit;
9. Other routine examinations are within the normal range or considered acceptable by the researchers.

Exclusion Criteria:

1. Recovery from major trauma (including surgery) within 4 weeks prior to study treatment;
2. Patients with systemic or locally severe infections, or other serious coexisting diseases;
3. Patients with allergies or allergies to any component of the imaging agent or antibody;
4. Patients who cannot perform PET/CT imaging scan;
5. Patients with abnormal immune function or who have recently used immunosuppressive or potentiating agents including various vaccines;
6. Patients with autoimmune diseases, including rheumatoid arthritis;
7. Inadequate control of arrhythmias, including atrial fibrillation;
8. Uncontrolled hypertension;
9. Syphilis, HBV, HCV, or HIV positive subjects;
10. Male and female subjects of reproductive age cannot take effective contraceptive measures;
11. Pregnant or lactating women;
12. Patients with a history of mental illness or related conditions;
13. Other subjects considered unsuitable by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Focal lesion of 89Zr-NY001 PET scanning in patients with fibronectin ED-B domain positive solid tumors. | 1 year
  Degree and localization of focal lesion compared with that of 18F-FDG PET scans and according to the expression of fibronectin ED-B domain will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi No. 4 People's Hospital, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No